CLINICAL TRIAL: NCT01174940
Title: A Study of Extracorporeal Photopheresis With UVADEX® in the Setting of a Standard Myeloablative Conditioning Regimen in Related or Unrelated Donor Hematopoietic Stem Cell Transplantation for the Prevention of Graft Versus Host Disease
Brief Title: Test Extracorporeal Photopheresis (ECP) Treatment Before/After Allogeneic Bone Marrow Transplant (BMT) or Peripheral Blood Stem Cell (PBSC) Transplant to Prevent Graft Versus Host Disease
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: Mallinckrodt (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12047
Record Dates: First submitted 2010-07-27; First posted 2010-08-04 (Estimated); Last update posted 2017-01-09 (Estimated); Status verified 2017-01

CONDITIONS: Stem Cell Leukemia of Unclear Lineage; Graft Versus Host Disease
Keywords: myelogenous leukemia; lymphocytic leukemia; lymphoblastic leukemia; myelodysplastic syndrome; non-Hodgkin's lymphoma; Hodgkin's disease
MeSH Terms: conditions — Graft vs Host Disease; Leukemia, Myeloid; Leukemia, Lymphoid; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Myelodysplastic Syndromes; Lymphoma, Non-Hodgkin; Hodgkin Disease | interventions — Photopheresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Extracorporeal Photopheresis (Experimental): Patients will receive 2 ECP treatments on day -10 and day -8 and then for two consecutive days every two weeks starting from post engraftment (ANC > 500) up to day 90 (total of 10 treatments). This may be given as an outpatient procedure.
  Interventions: Drug: extracorporeal photopheresis

INTERVENTIONS:
Drug: extracorporeal photopheresis — Patients will receive 2 ECP treatments prior to the commencement of the high dose chemotherapy and then for two consecutive days every two weeks starting from post engraftment (ANC > 500) up to day 90 (total of 10 treatments). This may be given as an outpatient procedure.
  The dose of UVADEX® used to inoculate these cells will be calculated based on the treatment volume collected during the plasma/buffy coat collection process, using the following formula:
  Treatment Volume in mL X 0.017 of UVADEX® (20 mcg/ml) required for administration into the recirculation bag = Amount of UVADEX® (in mLs) required for administration into the recirculation bag.
  After the cells are inoculated with UVADEX®, the buffy coat/plasma suspension is irradiated with ultraviolet-A light and then re-infused back into the patient.
  Other Names: UVAR; UVAR XTS

SUMMARY:
To study the effect of ECP with Uvadex® in conjunction with a standard myeloablative conditioning regimen on the incidence of acute and chronic GvHD in patients undergoing an allogeneic related or unrelated BMT or PBSC transplant, for treatment of hematologic or lymphoproliferative malignancies.

DETAILED DESCRIPTION:
This study is to test the concept that using ECP treatment prior to and after an allogeneic bone marrow transplant (BMT) or peripheral blood stem cell (PBSC) transplant will prevent the development of GvHD. This study is not designed to detect a specific treatment effect. However, some statements about the outcome of the study are possible. A sample size of n = 21 patients could detect a statistically significant difference between the expected rate of GvHD in an untreated population, 60%, and our hypothesized rate, 30%, for the matched-unrelated recipients. This calculation is based on a one-sample, two-sided chi-square test at the 5% level of significance with 80% power.

Patients will receive ECP from day -10 and day -8 before transplant and then from day of engraftment absolute neutrophil count (ANC>500) until day 90 after transplant. Patients who enter the study will receive a BMT or PBSC transplant from a donor who is matched unrelated (8/10 to 10/10 match). Rates of acute GvHD and chronic GvHD that occur in patients are 50-70% for the matched-unrelated donor transplant.

The choice of sample size is 21 patients. The analysis will determine if there are favorable trends for a treatment effect. Comparison on survival, and rates of acute and chronic GvHD will be made with historical controls who have undergone similar myeloablative transplant from an unrelated donor.

ELIGIBILITY:
Inclusion Criteria:

* Patients are eligible if they have a diagnosis of one of the following hematologic or lymphoproliferative malignancies for which a treatment option would be an allogeneic BMT or PBSC transplant:

  * acute myelogenous leukemia
  * chronic myelogenous leukemia
  * acute lymphocytic/blastic leukemia
  * chronic lymphocytic leukemia
  * myelodysplastic syndrome
  * non-Hodgkin's lymphoma (expected survival > 60 days)
  * Hodgkin's disease (expected survival > 60 days)
* Patients who are candidates for a standard allogeneic BMT or patients who are candidates for a standard allogeneic PBSC transplant.
* Patients must have a suitable HLA- molecular matched (8/10 or more) related or unrelated donor.
* Patients must be physically and psychologically capable of undergoing a BMT or PBSC transplant and the attendant period of strict isolation.
* Patients must test negative for human immunodeficiency virus (HIV).
* Patients must present no evidence of active ongoing infection.
* Patients must have adequate renal, hepatic, pulmonary, and cardiac function to enable the patient to tolerate the extracorporeal volume shifts associated with ECP, as determined by the physician's clinical judgment.
* Platelets ≥ 20,000/cmm.
* Patients ≥ 18 years of age.
* Weight ≥ 40 kg (88 lb).
* Systolic Blood Pressure ≥ 90 mm Hg after the patient has been in a sitting position for five minutes.
* Women of childbearing potential must agree to use a reliable method of birth control for the duration of the study.
* Patients must be willing to comply with all study procedures.
* Signed and dated informed consent must be obtained prior to conducting any study procedures. The parent or legal guardian of a minor must also provide written informed consent.

Exclusion Criteria

* Patients who have received a prior allogeneic BMT or PBSC transplant.
* Hypersensitivity or allergy to psoralen (methoxsalen).
* Contraindication to radiation, cyclophosphamide, CSA, Busulphan or MTX.
* Hypersensitivity or allergy to both heparin and citrate products. (If hypersensitive or allergic to only one of these two products, exclusion does not apply if the other product is strictly used for the patient.)
* Patients whose treatment requires donor lymphocyte infusion up to day 100 post-transplant.
* Participation in another clinical trial for prevention of GvHD within 7 days prior to patient enrollment or concurrent participation in any other clinical study.
* Active gastrointestinal bleeding.
* Females who are pregnant or lactating.
* Previous treatment with ECP.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2010-06; Primary Completion 2014-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Presence/absence of grade II-IV acute Graft versus Host Disease (aGVHD) | 100 days after transplant
  The primary efficacy variable is the presence/absence of grade II-IV acute GvHD within the first 100 days after transplantation

SECONDARY OUTCOMES:
proportion of patients who develop chronic Graft versus Host Disease (cGVHD) and experience relapse of primary disease. | 365 days after transplantation
  These secondary efficacy variables for a patient are dichotomous:
  * the development of cGvHD during 365 days after transplantation (and which body sites are involved)
  * the relapse of primary disease (hematologic or lymphoproliferative malignancy)
  * the grade of aGvHD
  * the involved sites of cGvHD

CONTACTS AND LOCATIONS:
Overall Officials: Sunil Abhyankar, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States